CLINICAL TRIAL: NCT03735043
Title: Continuous Non-invasive Cardiac Output, an Evaluation of ccNexfin© in a Pregnant Population
Brief Title: Cardiac Output Monitoring by ccNexfin© in Pregnant Women
Acronym: CoNex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017_54; 2018-A01089-46 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2018-09-18; First posted 2018-11-08 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Pregnancy
Keywords: Pregnancy; ccNexfin©; cardiac output; hemodynamic; non-invasive monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ccNexfin © (Experimental)
  Interventions: Device: cardiac output by ccNexfin ©

INTERVENTIONS:
Device: cardiac output by ccNexfin © — Measurement of cardiac output by ccNexfin © comparatively to transthoracic echocardiography Subjects participating to the study will be simultaneously measured for cardiac output by ccNexfin © and transthoracic echocardiography. Echocardiographic measurements of cardiac output will be blinded to values measured by ccNexfin ©. For each participant, a first measurement of cardiac output will be performed in the supine position and then after 1 minute of strict left lateral position.

SUMMARY:
Variations of cardiac output are frequent in pregnant women during obstetrical procedures, and may participate to poor foetal outcomes through decrease of uteroplacental bloodflow. Thus, monitoring maternal cardiac output appears of major interest, as it would open the way to early initiation of hemodynamic supportive management.

The ccNexfin© is a non-invasive hemodynamic monitoring device, whose relevance for continuous monitoring of cardiac output has been reported in a non-pregnant population.

The hypothesis is that ccNexfin© gives acceptable measurement of maternal cardiac output in pregnant women.

ELIGIBILITY:
Inclusion Criteria

* Pregnancy > 32 weeks of amenorrhea
* Informed consent to participate to the study
* Health insurance

Exclusion Criteria:

* Poor echogenicity for Transthoracic echocardiography
* Cardiopathy
* Difficulties to move
* Necessity of strict supine or lateral position
* Impossibility to receive information or to give inform consent to participate to the study Refusal to sign inform consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant
Enrollment: 100 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Intra-class correlation coefficient between values of supine position cardiac output evaluated simultaneously by transthoracic echocardiography (measured in liters / minute) and ccNexfin © (measured in liters / minute) | 1 minute after positioning in supine position

SECONDARY OUTCOMES:
Cohen's Kappa coefficient between changes in maternal ejection volume observed from supine position to left lateral position, evaluated by transthoracic echocardiography (in %) and ccNexfin © (in %) respectively, at the 10% threshold of variation | Maternal ejection volume in supine position: 1 minute after positioning in supine position Maternal ejection volume in left lateral position: 1 minute after positioning in left lateral position
Cohen's Kappa coefficient between changes in maternal cardiac output observed from supine position to left lateral position, assessed by transthoracic echocardiography (in %) and ccNexfin © (in %) respectively, at the 15% threshold of variation | Maternal cardiac output in supine position: 1 minute after positioning in supine position Maternal cardiac output in left lateral position: 1 minute after positioning in left lateral position
Intra-class correlation coefficient between left lateral position cardiac output values assessed simultaneously by transthoracic echocardiography (measured in liters / minute) and ccNexfin © (measured in liters / minute) | 1 minute after positioning in left lateral position
Pearson correlation coefficient between values of supine position maternal cardiac output evaluated by transthoracic echocardiography (measured in liters / minute) and ccNexfin © (measured in liters / minute), respectively | 1 minute after positioning in supine position
Pearson correlation coefficient between values of left lateral position maternal cardiac output evaluated by transthoracic echocardiography (measured in liters / minute) and ccNexfin © (measured in liters / minute), respectively | 1 minute after positioning in left lateral position

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre GAUDET, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital coeur poumon, CHU, Lille, France

REFERENCES:
- [Derived] Bonnin P, Constans B, Duhamel A, Kyheng M, Ducloy-Bouthors AS, Estevez MG, Tavernier B, Gaudet A. Accuracy and trending ability of finger plethysmographic cardiac output monitoring in late pregnancy. Can J Anaesth. 2022 Nov;69(11):1340-1348. doi: 10.1007/s12630-022-02297-y. Epub 2022 Aug 4. PMID 35927539